CLINICAL TRIAL: NCT06408389
Title: From Oocyte to Embryo: Analysis of Mechanics of Human Pre Implantation Development
Brief Title: Mechanics of Human Pre Implantation Development
Acronym: MECANEMB
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Collège de France (Unknown); Institut Curie (Other); Centre National de la Recherche Scientifique, France (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210563
Record Dates: First submitted 2021-11-16; First posted 2024-05-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infertility
Keywords: In vitro fertilization; embryo; human time lapse; pregnancy; delivery; machine learning
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The time-lapse is a closed tri-gas incubator of the latest generation that provides optimal and stable culture conditions for the culture of embryos in In Vitro Fertilization (IVF). The integration of a camera within this incubator allows for continuous image capture, thus facilitating the monitoring of the entire embryonic development, from the day of fertilization to the moment of transfer into the uterus.

The contribution of the time-lapse system allows an evaluation of the embryos not only by their morphology, but also by their cell division kinetics, both being direct markers of cell mechanics. Together, these morpho-kinetic data finally allow for the best identification of embryos with greater implantation potential. Time-lapse imaging represents a further step towards an objective assessment of the embryo, but inter- and intra-embryologist variations in annotations partly compromise this objectivity. In addition, many decision algorithms based on the evaluation of morpho-kinetic parameters have been developed, but the lack of reproducibility from one Assisted Reproductive Technology (ART) center to another is a hindrance to the generalization of any particular algorithm. The aim of this retrospective study is to determine morpho-kinetic factors predictive of implantation using machine learning and to link these factors to human embryo mechanistic properties.

DETAILED DESCRIPTION:
The time-lapse is a closed tri-gas incubator of the latest generation that provides optimal and stable culture conditions for the culture of embryos in In Vitro Fertilization (IVF). The integration of a camera within this incubator allows for continuous image capture, thus facilitating the monitoring of the entire embryonic development, from the day of fertilization to the moment of transfer into the uterus.

The contribution of the time-lapse system allows an evaluation of the embryos not only by their morphology, but also by their cell division kinetics, both being direct markers of cell mechanics. Together, these morpho-kinetic data finally allow for the best identification of embryos with greater implantation potential. Time-lapse imaging represents a further step towards an objective assessment of the embryo, but inter- and intra-embryologist variations in annotations partly compromise this objectivity. In addition, many decision algorithms based on the evaluation of morpho-kinetic parameters have been developed, but the lack of reproducibility from one Assisted Reproductive Technology (ART) center to another is a hindrance to the generalization of any particular algorithm.

Machine learning is one of the main methods of data analysis that could define algorithms that are unbiased, more robust and applicable to all centers. But the optimal algorithm is not yet defined. Recently, an artificial intelligence approach applied to a large collection of time-lapse embryo images was developed to determine the embryo with the highest grade of evolution, with an AUC> 0.98. Using clinical data, the authors created a decision tree to integrate embryo quality and female age and identify the chances of pregnancy. However, this approach did not take into account the whole kinetics of development, focusing on certain particular stages, nor the influence of parental and extrinsic factors other than age.

The aim of this retrospective study is to determine morpho-kinetic factors predictive of implantation and embryo development in IVF/ICSI using machine learning algorithms and relate these morpho-kinetic factors to the mechanical characteristics of cells.

ELIGIBILITY:
Inclusion Criteria:

* Couples enrolled in an IVF process and with embryos cultured in time-lapse
* Couples informed non opposed to research

Exclusion Criteria:

* Couples opposed to research
* Couples under curator or tutorship
* Couples under state xxx

Ages: 18 Years to 43 Years | Sex: All
Age Groups: Adult
Study Population: Couples enrolled in an IVF process (conventional IVF or with sperm micro-injection (ICSI))
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Prediction of embryo implantation by the machine learning algorithm from embryo morphokinetic parameters and patient health data. | 2 years
  The algorithm outcome will be evaluated retrospectively on human embryos which have been transferred, for which we know whether its implantation was successful and led to birth. Using embryo morphokinetic and health patient data, we will predict a probability of implantion and compare its value (<0.5: no implantation or >0.5: implantation) to the true result of the embryo transfer (no implantation or implantation). This will allow us to evaluate the potential of the algorithm to support clinical decision-making in the future.

SECONDARY OUTCOMES:
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Age (years) : female / male
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Weight (kg) : female / male
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Height (cm) : female / male
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Weight and height combined for BMI (kg/M2) : female / male
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : Day-3 FSH (IU/l)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : Day-3 LH (IU/l)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : Day-3 Estradiol (pg/ml)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : Day-3 AMH (ng/ml)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : Day-3 Antral Follicular count
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : cause of infertility (endometriosis (yes/no))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : cause of infertility (tubal (yes/no))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Female : cause of infertility (diminished ovarian reserve (yes/no))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : sperm parameters (volume (ml))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : sperm parameters (concentration (10^6/ml))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : sperm parameters (progressive mobility (%))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : sperm parameters (vitality (%))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : sperm parameters (normal form (%))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : FSH (IU/l)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : LH (IU/l)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : total testosterone (ng/ml)
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  caryotype : Female/male
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : cause of male infertility (obstructive azoospermia (yes/no))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : cause of male infertility (non-obstructive azoospermia (yes/no))
Link between couples' parameters and embryo morpho-kinetics | 3 years
  Identify statistical links between parental or extrinsic factors (linked to the attempt) and morpho-kinetic parameters :
  Male : cause of male infertility (oligoasthenoteratospermia (yes/no))
Statistical correlation between embryo implantation prediction and morphokinetic parameters | 3 years
  The machine learning algorithm (neural network) trained for the primary outcome will be used to quantify the average percentage contributed by each morphokinetic parameter in the prediction of implantation success or failure ("explainable artificial intelligence"). This will allow us to determine what morphokinetic parameters influence the most positively or negatively the prediction of implantation.
Embryo reconstruction in 3D | 3 years
  Develop an automatic method for reconstructing the morphology of embryos in 3 dimensions from 2-dimensional images in transmitted light (Geri incubator or Embryoscope type)
Software developing | 3 years
  Develop decision support software for the benefit of embryologists as part of an ART attempt

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PATRAT, MD, PhD, Principal Investigator — AP-HP (Professor in Medicine faculty and Hospital practitioner (APHP.centre - Université de Paris, site Cochin); Jean-Léon MAITRE, PhD, Study Director — Institut Curie CNRS UMR3215 INSERM U934; Hervé TURLIER, Study Director — Collège de France, CIRB CNRS UMR7241

IPD SHARING:
Plan to Share IPD: No